CLINICAL TRIAL: NCT02682303
Title: Effect of Elastic Bandage on Measurements of Balance in Subjects With Chronic Ankle Instability: a Randomized Clinical Trial
Brief Title: Effect of Elastic Bandage on Balance in Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05/14
Record Dates: First submitted 2016-01-28; First posted 2016-02-15 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Ankle Sprain
Keywords: Adhesive elastic bandaging; balance; posturography
MeSH Terms: conditions — Ankle Injuries | interventions — Compression Bandages

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- elastic bandage (Experimental): In this study, Idealplast C® (6cm*2.5m) was used.
  Interventions: Device: Elastic Bandage (Idealplast C®)
- Non-standardized tape (NST) (Placebo Comparator): In the NST group, Pretape Cramer® (100% cotton, 1.25cm*10m) was used.
  Interventions: Device: Pretape cramer® (non standarized tape)

INTERVENTIONS:
Device: Elastic Bandage (Idealplast C®) — Elastic bandage
  One anchor strip is applied around the ankle with no tension applied to the tape to avoid restricting blood flow. A supporting stirrup strap is applied from the inside of the ankle, under the heel with no tension up to this point. As the tape is passed up the outside of the ankle tension is applied to the tape with the foot in slight dorsiflexion and secured to the anchor strap (black arrow).
  For heel lock, a second strip is applied on the outside of the ankle, taken across the front of the ankle and just above the bony part on the inside of the ankle and back towards the heel (red arrow). Then taken around and under the heel back the way you have just come and around the front of the ankle (orange arrow). The tape then passes above the bony part of the ankle on the outside and diagonally towards the heel, across to the inside of the ankle then around the top to finish
  Arms: elastic bandage
Device: Pretape cramer® (non standarized tape) — Pretape cramer® was used.
  The individual is in supine position keeping the foot and ankle in a neutral position.
  The strip (I) is applied with not stretch in the outside of the leg just above the ankle, and then the rest of the strip is applied on the outside of the ankle and under the heel.
  This is the only intervention carried out in this group.
  Arms: Non-standardized tape (NST)

SUMMARY:
Purpose: To report the immediate and prolonged (one week) effects of elastic bandage on balance control in subjects with chronic ankle instability.

Material and methods: Twenty-eight individuals successfully completed the study protocol, of whom 14 were randomly assigned to the elastic bandage group (7 men, 7 women) and 14 were assigned to the non-standardized tape group ( 9 men, 5 women). To objectively measure postural sway we used computerized dynamic posturography with Sensory Organization Test and Unilateral Stance test. We analyzed the following Sensory Organization Test parameters: the composite Sensory Organization Test score, the composite Sensory Organization Test strategy and the Sensory Organization Test condition 2 and its strategy. In addition, we studied the centre of gravity sway velocity with open eyes and close eyes during the US test.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Chronic Ankle Instability

Exclusion Criteria:

Neurologic disease Vestibular disease

Ages: 18 Years to 28 Years | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Balance using a computerized dynamic posturography test: the sensory organization test | 7 days
  The CDP device employed in this study was Smart Equitest® version 8.2 (NeuroCom International Inc., Clackamas, OR, USA). Posturography analysis was conducted using the SOT. This test assesses postural control through the use of external stimuli on the visual and proprioceptive system.
  Participants were instructed to stand on the force-plate facing the visual surround. A safety harness was fixed to prevent injury from falls. Their bare feet position on force-plates was adjusted according to the height of the patient, as marked on the equipment. Subjects had to maintain their COG stable in 3 consecutive series of 20s duration for each of the 6 conditions in the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Francisco Molina Rueda. Avda. de Atenas. s/n., Alcorcón, Madrid, Spain

REFERENCES:
- See also: University — http://www.urjc.es